CLINICAL TRIAL: NCT02477306
Title: Comparative Open-label,Randomized, Fasting, Single Dose, Two-way Crossover Bioequivalence Study of Rabeprazole From Idiazole 20mg DR Tabs (GSK, Egypt) and PARIET 20 mg DR Tabs (JANSSEN, EGYPT)
Brief Title: A Bioequivalence Study of Rabeprazole From Idiazole 20mg DR Tabs (GSK, Egypt) and PARIET 20 mg DR Tabs (JANSSEN, EGYPT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GRC1/14/516GSKRABFST
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): 60 subjects will receive a single oral dose of idiazole 20mg DR tabs under fasting condition in one period. And the subjects will receive a single dose of PARIET 20 mg DR tabs under fasting condition in the second period. A 7 days washout interval is in between the 2 periods
  Interventions: Drug: Idiazole 20mg DR tabs; Drug: PARIET 20 mg DR tabs

INTERVENTIONS:
Drug: Idiazole 20mg DR tabs — Delayed release tablets containing 20 mg of rabeprazole
Drug: PARIET 20 mg DR tabs — Orally administered, delayed-release, enteric-coated tablets containing 20 mg of rabeprazole sodium.

SUMMARY:
Comparative randomized, single dose, two-way crossover open-label study to determine the bioequivalence of Rabeprazole from Idiazole 20mg DR tabs (GSK, Egypt)and PARIET 20 mg DR tabs (JANSSEN, EGYPT) after a single oral dose administration of each to healthy adults under fasting conditions.

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e. The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects whose values of BMI were outside the accepted normal ranges.
3. Female subjects who are pregnant, nursing or taking birth control pills.
4. Medical demographics with evidence of clinically significant deviation from normal medical condition.
5. Results of laboratory tests which are clinically significant.
6. Acute infection within one week preceding first study drug administration.
7. History of drug or alcohol abuse.
8. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
9. Subject is on a special diet (for example subject is vegetarian).
10. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
11. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
12. Subject has a history of severe diseases which have direct impact on the study.
13. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
14. Subject intends to be hospitalized within 6 weeks after first study drug administration.
15. Subjects who, through completion of this study, would have donated more than 500 ml of blood in 7 days, or 750 ml of blood in 30 days, 1000 ml in 90 days, 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Maximal measured plasma concentration (Cmax) | Up to 14 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected pre-dose and at 0.00, 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.33, 4.67, 5.0, 5.33, 5.67, 6.00, 8.00, 12.0 and 14.0 hours post dose, relative to dosing on Day 1 in each cross over period.
Area under the plasma concentration-time curve from time zero to the last measurable concentration (t) (AUC [0 to t]) | Up to 14 hours post dose in each treatment period
  (AUC [0 to t]) will be calculated by the linear trapezoidal method.
Area Under the plasma concentration-time curve from time zero to infinity (AUC [0 to infinity]) | Up to 14 hours post dose in each treatment period
  AUC (0 to infinity) will be calculated as the sum of the AUC (0 to t) plus the ratio of the last measurable plasma concentration to the elimination rate constant

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (tmax) | Up to 14 hours post dose in each treatment period
  If the Tmax occurs at more than time point, then tmax will be considered for the first occurrence.
Apparent first-order elimination or terminal rate constant (K¬e) | Up to 14 hours post dose in each treatment period
  K¬e will be calculated from a semi-log plot of the plasma concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations
Terminal half life (t1/2e) | Up to 14 hours post dose in each treatment period
  The elimination or terminal half-life will be calculated as 0.693/ Ke

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

REFERENCES:
- See also: International conference of Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline Q2B. Guidelines for Validation of Analytical Procedures: Methodology. November, 1996 — http://www.pharmaweb.net/pwmirror/pw9/ifpma/ICH1.html